CLINICAL TRIAL: NCT00505037
Title: A Phase 2, Randomized, Double-blind-placebo-controlled and Open-label-Sevelamer Hydrochloride-controlled, Dose-ranging Study for ASP1585 in Patients With Chronic Kidney Disease(CKD) and Hyperphosphatemia on Hemodialysis
Brief Title: A Phase 2 Study of ASP1585 in Chronic Kidney Disease Patients With Hyperphosphatemia on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1585-CL-0002
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: ASP1585; Renal Dialysis; Chronic Kidney Disease; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ASP1585 dose #1 (Experimental)
  Interventions: Drug: ASP1585
- ASP1585 dose #2 (Experimental)
  Interventions: Drug: ASP1585
- ASP1585 dose #3 (Experimental)
  Interventions: Drug: ASP1585
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Sevelamer hydrochloride (Active Comparator)
  Interventions: Drug: Sevelamer hydrochloride

INTERVENTIONS:
Drug: ASP1585 — Oral
  Arms: ASP1585 dose #1; ASP1585 dose #2; ASP1585 dose #3
Drug: Placebo — Oral
  Arms: Placebo
Drug: Sevelamer hydrochloride — Oral
  Arms: Sevelamer hydrochloride

SUMMARY:
To evaluate the superiority to placebo, dose-responsibility and safety.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind placebo-controlled and open label sevelamer hydrochloride-controlled, dose-ranging study in CKD patients with hyperphosphatemia on hemodialysis. Patients will be randomly allocated to one of the five treatment groups (ASP1585: 3 dose, placebo, Sevelamer hydrochloride) and advance to the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Stable CKD patients who are currently on hemodialysis three times a week for at least 12 weeks prior to the acquisition of informed consent
* Patients on stable dose(s) of phosphate binder(s) for at least 28 days prior to the acquisition of informed consent.
* Patients on stable dose(s) of Vitamin D or calcitonin agent for at least 28 days prior to the acquisition of informed consent, in case patients are treated by those agents

Exclusion Criteria:

* History of major gastrointestinal surgery, or swallowing disorders, bowel obstruction, hemorrhagic gastrointestinal lesion
* Continuous severe constipation/diarrhea.
* History of parathyroid intervention [parathyroidectomy（PTx），percutaneous ethanol injection therapy（PEIT）etc.] within 1 year of the acquisition of informed consent
* Diet restriction such as fasting and/or excessive dieting
* Uncontrolled hypertension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in serum phosphorus | 4 weeks

SECONDARY OUTCOMES:
Change in serum phosphorus level by time | Up to 4 weeks
Percent of patients meeting the target range of serum phosphorus (3.5-6.0 mg/dL) and achieving time | 4 Weeks
Change in corrected serum Ca level | 4 weeks
Change in Ca×P | 4 weeks
Change in intact PTH | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chugoku
  - Chūbu
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Akizawa T, Origasa H, Kameoka C, Kaneko Y, Kanoh H. Dose-finding study of bixalomer in patients with chronic kidney disease on hemodialysis with hyperphosphatemia: a double-blind, randomized, placebo-controlled and sevelamer hydrochloride-controlled open-label, parallel group study. Ther Apher Dial. 2014 Jun;18 Suppl 2:24-32. doi: 10.1111/1744-9987.12202. PMID 24975892